CLINICAL TRIAL: NCT02658240
Title: Ultrasound-guided Fascia Iliaca Compartment Block Versus Periarticular Infiltration for Pain Management After Total Hip Arthroplasty: A Randomized Controlled Trial
Brief Title: Ultrasound-guided Fascia Iliaca Compartment Block Versus Periarticular Infiltration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Irina Gasanova, Associate Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STU 122015-022
Record Dates: First submitted 2016-01-14; First posted 2016-01-18 (Estimated); Results first posted 2018-11-29 (Actual); Last update posted 2018-11-29 (Actual); Status verified 2018-11

CONDITIONS: Postoperative Pain
Keywords: Nerve block; Periarticular infiltration; Ropivacaine; Pain
MeSH Terms: conditions — Pain, Postoperative; Pain | interventions — Ropivacaine; Epinephrine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Compartment Block (Active Comparator): Fascia iliaca compartment block (FICB) with ropivacaine and epinephrine after surgery
  Interventions: Drug: Ropivacaine; Drug: Epinephrine
- Infiltration (Active Comparator): Periarticular infiltration with ropivacaine and epinephrine prior to closing the incision
  Interventions: Drug: Ropivacaine; Drug: Epinephrine

INTERVENTIONS:
Drug: Ropivacaine — Ropivacaine 300 mg and 0.5 mg epinephrine diluted to 60 mL
Drug: Epinephrine — 0.5 mg epinephrine
  Other Names: Adrenaline

SUMMARY:
This randomized, controlled, observer-blinded study clinical trial was designed to evaluate ultrasound-guided fascia iliaca compartment block with ropivacaine and periarticular infiltration with ropivacaine for postoperative pain management after total hip arthroplasty.

DETAILED DESCRIPTION:
Despite substantial advances in our understanding of the pathophysiology of pain and availability of newer analgesic techniques, postoperative pain is not always effectively treated. Optimal pain management technique balances pain relief with concerns about safety and adverse effects associated with analgesic techniques. Currently, postoperative pain is commonly treated with systemic opioids, which are associated with numerous adverse effects including nausea and vomiting, dizziness, drowsiness, pruritus, urinary retention, and respiratory depression. Use of regional and local anesthesia has been shown to reduce opioid requirements and opioid-related side effects.

Patients undergoing total hip arthroplasty (THA) (n=60) at Parkland and UT Southwestern Medical Center Hospitals will be randomized into one of two groups to receive either ultrasound-guided fascia iliaca compartment block (FICB) with ropivacaine 300 mg and 0.5 mg epinephrine (Group 1) or periarticular infiltration ropivacaine 300 mg and 0.5 mg epinephrine total (Group 2) for postoperative pain management. The remaining aspect of perioperative care, including the anesthetic technique (i.e., spinal anesthetic), pre- and postoperative care will be standardized and will be similar for all patients. The duration of the involvement in the study will be until 48 hours postoperatively.

Patients in Group 1 will receive ultrasound-guided FICB after surgery. Patients in Group 2 will receive ropivacaine via periarticular infiltration prior to closing the incision.

The postoperative analgesia will be documented using the visual analog score (0=no pain, 10=worst pain). In addition, total opioid dose over the 48-h study period will be documented. Postoperative nausea will be measured using a categorical scoring system (none=0, mild=1, moderate=2, severe=3) and episodes of vomiting will be documented. Rescue antiemetics will be given to any patient who complains of nausea and/or vomiting. All variables will be assessed at 2, 6, 12, 24, and 48 hours, postoperatively by an investigator blinded to group allocation.

ELIGIBILITY:
Inclusion Criteria:

* Female ASA physical status 1-3 scheduled for total hip arthroplasty
* Age 18-80 years old
* Able to participate personally or by legal representative in informed consent in English or Spanish

Exclusion Criteria:

* History of relevant drug allergy
* Age less than 18 or greater than 80 years
* Chronic opioid use or drug abuse
* Significant psychiatric disturbance
* Inability to understand the study protocol
* Refusal to provide written consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-04-05 (Actual); Primary Completion 2017-11-13 (Actual); Study Completion 2017-12-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Irina Gasanova, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UTSW Parkland Health Hospital System, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gasanova I, Alexander JC, Estrera K, Wells J, Sunna M, Minhajuddin A, Joshi GP. Ultrasound-guided suprainguinal fascia iliaca compartment block versus periarticular infiltration for pain management after total hip arthroplasty: a randomized controlled trial. Reg Anesth Pain Med. 2019 Feb;44(2):206-211. doi: 10.1136/rapm-2018-000016. PMID 30700615

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Compartment Block | Infiltration
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Compartment Block | Infiltration | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.2 (13.6) | 59.0 (11.2) | 57.6 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 18 | 36
  Male | 12 | 12 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 11 | 23
  Not Hispanic or Latino | 18 | 19 | 37
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30 | 30 | 60
Preoperative Pain Score at Rest [Median (Inter-Quartile Range); unit: units on a scale] — The Visual Analog Pain Score (VAS) on the scale of 10 (0= No pain, 10= Worst pain) at preoperatively
  units on a scale | 3 [0 to 4] | 4 [3 to 6] | 4 [2 to 6]
Preoperative Pain Score with Cough [Median (Inter-Quartile Range); unit: units on a scale] — The Visual Analog Pain Score (VAS) with cough on the scale of 10 (0= No pain, 10= Worst pain) preoperatively
  units on a scale | 4 [3 to 5] | 8 [7 to 10] | 8 [6.75 to 10]

OUTCOME MEASURES:

1. Primary Outcome: Postoperative Pain Score at Resting
Description: The Visual Analog Pain Score (VAS) at resting on the scale of 10 (0= No pain, 10= Worst pain) at 48 hours postoperatively
Time Frame: Postoperative 48 hours
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Compartment Block | Infiltration
Number analyzed (Participants) | 30 | 30
units on a scale | 1 [0 to 2] | 2 [1 to 2]
Statistical Analysis 1: Comparison: Compartment Block vs Infiltration; The study was powered to detect a mean difference of 1.5 in pain scores in favor of patients undergoing SFICB procedure assuming a standard deviation of 2.5. With a two sided alpha level of 0.05, a total of 52 patients would be needed to have 80% power using a repeated measures ANOVA F test with 6 observations on each subject. Correlation on the repeat observations was assumed to be 0.5. Assuming a 14% loss to follow-up, 60 patients were enrolled at 1:1 ratio; Test type: Superiority; p = 0.05, ANOVA

2. Primary Outcome: Postoperative Pain Score With Movement
Description: The Visual Analog Pain Score (VAS) with movement on the scale of 10 (0= No pain, 10= Worst pain) at 48 hours postoperatively
Time Frame: Postoperative 48 hours
Measure: Mean (Inter-Quartile Range); unit: units on a scale
Arm/Group | Compartment Block | Infiltration
Number analyzed (Participants) | 30 | 30
units on a scale | 3 [2 to 4] | 4 [3 to 5]
Statistical Analysis 1: Comparison: Compartment Block vs Infiltration; Test type: Superiority; p = 0.05, ANOVA

3. Secondary Outcome: Oral Morphine Equivalents of Postoperative Opioid Requirements for 48 Hours
Description: Total amounts of postoperative opioid requirements for 48 hours postoperatively
Time Frame: Postoperative 48 hours
Measure: Mean (Standard Deviation); unit: Oral Morphine Equivalent (mg)
Arm/Group | Compartment Block | Infiltration
Number analyzed (Participants) | 30 | 30
Oral Morphine Equivalent (mg) | 101.0 (29.5) | 115.6 (46)
Statistical Analysis 1: Comparison: Compartment Block vs Infiltration; Test type: Superiority; p = 0.149, t-test, 2 sided

4. Secondary Outcome: The Time to Ambulation
Description: The time to ambulation during 48 hours postoperative period
Time Frame: Postoperative 48 hours
Measure: Median (Inter-Quartile Range); unit: Hours
Arm/Group | Compartment Block | Infiltration
Number analyzed (Participants) | 30 | 30
Hours | 21.3 [19 to 23.5] | 22 [19.5 to 24]
Statistical Analysis 1: Comparison: Compartment Block vs Infiltration; Test type: Superiority; p = 0.584, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected during 48 hours postoperatively.
Arm/Group | Compartment Block | Infiltration
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-04-01): https://cdn.clinicaltrials.gov/large-docs/40/NCT02658240/Prot_SAP_000.pdf